CLINICAL TRIAL: NCT04604756
Title: Losartan Effects on the Social Reward in Humans
Brief Title: The Effects of Losartan on Social Reward
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-72
Record Dates: First submitted 2020-10-09; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Healthy
Keywords: Losartan; Social reward
MeSH Terms: interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Losartan group (Experimental): Drug: Losartan
  Interventions: Drug: Losartan
- Placebo group (Placebo Comparator): Drug: Placebo Oral Tablet
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Losartan — administration of losartan (50 mg) (oral)
  Other Names: Cozaar Oral Tablet
  Arms: Losartan group
Drug: Placebo Oral Tablet — administration of placebo (oral)
  Arms: Placebo group

SUMMARY:
The aim of the study is to investigate the effect of losartan (50mg, single dose) on social reward

DETAILED DESCRIPTION:
In a double-blind, between-subject, placebo-controlled design the effects of a single dose of losartan (50mg) on social reward in healthy participants will be examined. 90 minutes after subjects administrate 50mg losartan or placebo, participants will undergo a social incentive delay task. Neural activity will be assessed by the acquisition of functional magnetic resonance imaging (fMRI) data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* history of head injury
* medical or psychiatric illness
* hypertension

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Losartan effects on neural activity as assessed by blood oxygenation dependent (BOLD) fMRI during the anticipation of social feedback. | 90 minutes to 105 minutes after treatment
  The social incentive delay task provides subjects with trial-wise feedback on their performance (as assessed by reaction time). Neural activity will be measured by functional magnetic resonance imaging (fMRI). To examine effects of treatment during the anticipation of social feedback fMRI-based neural indices during the anticipation period will be compared between the losartan and the placebo treated group using a Generalized Linear Model approach. The analysis will focus on brain systems that play an important role in the anticipation of reward and punishment (prefrontal cortex and subcortical regions, including the striatum)
Losartan effects on neural activity as assessed by blood oxygenation dependent (BOLD) fMRI during the consummation of social feedback. | 90 minutes to 105 minutes after treatment
  The social incentive delay task provides subjects with trial-wise feedback on their performance (as assessed by reaction time). Following each trial the feedback will be indicated by positive and negative social stimuli. Neural activity will be measured by functional magnetic resonance imaging (fMRI). To examine effects of treatment during the consummation of social feedback fMRI-based neural indices during the presentation of the feedback will be compared between the losartan and the placebo treated group using a Generalized Linear Model approach. The analysis will focus on brain systems that play an important role in reward and punishment (prefrontal cortex and subcortical regions, including the striatum)

SECONDARY OUTCOMES:
Effects of Losartan on arousal ratings of the stimuli presented during the fMRI-paradigm as assessed by 1-9 Likert scales | 150 minutes to 160 minutes after treatment
  Following the fMRI assessment participants will be asked to rate the arousal of the stimuli presented during fMRI. Arousal will be assessed on 1-9 Likert rating scales. To examine effects of treatment on arousal ratings the losartan and placebo groups will be compared using Generalized Linear Model approach.
Effects of Losartan on valence ratings of the stimuli presented during the fMRI-paradigm as assessed by 1-9 Likert scales | 150 minutes to 160 minutes after treatment
  Following the fMRI assessment participants will be asked to rate the valence of the stimuli presented during fMRI. Valence will be assessed on 1-9 Likert rating scales. To examine effects of treatment on valence ratings the losartan and placebo groups will be compared using Generalized Linear Model approach.
Effects of Losartan on intensity ratings of the stimuli presented during the fMRI-paradigm as assessed by 1-9 Likert scales | 150 minutes to 160 minutes after treatment
  Following the fMRI assessment participants will be asked to rate the intensity of the stimuli presented during fMRI. Intensity will be assessed on 1-9 Likert rating scales. To examine effects of treatment on intensity ratings the losartan and placebo groups will be compared using Generalized Linear Model approach.
Effects of Losartan on likeability ratings of the stimuli presented during the fMRI-paradigm as assessed by 1-9 Likert scales | 150 minutes to 160 minutes after treatment
  Following the fMRI assessment participants will be asked to rate the likeability of the stimuli presented during fMRI. Likeability will be assessed on 1-9 Likert rating scales. To examine effects of treatment on likeability ratings the losartan and placebo groups will be compared using Generalized Linear Model approach.
Effects of Losartan on dislikeability ratings of the stimuli presented during the fMRI-paradigm as assessed by 1-9 Likert scales | 150 minutes to 160 minutes after treatment
  Following the fMRI assessment participants will be asked to rate the dislikeability of the stimuli presented during fMRI. Dislikeability will be assessed on 1-9 Likert rating scales. To examine effects of treatment on dislikeability ratings the losartan and placebo groups will be compared using Generalized Linear Model approach.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Becker, PhD, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No